CLINICAL TRIAL: NCT06571539
Title: High-accuracy Augmented Reality Guidance for Intracranial Drain Placement Using a Standalone Head-worn Navigation System
Brief Title: Augmented Reality-Assisted Neurosurgical Drain Placement
Acronym: ARANED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other); Imec (Industry); Orsi Academy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UZB-ARANED-1
Record Dates: First submitted 2024-07-31; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2018-11

CONDITIONS: Intracranial Hypertension
Keywords: Augmented reality; Neuronavigation; Computer-assisted surgery; Ventricular drain placement; Ventriculostomy
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective clinical pilot study with the goal to assess feasibility, safety and clinical performance of high-accuracy AR-guided EVD placement using a standalone head-worn navigation system in critical care settings at the Universitair Ziekenhuis Brussel over the course of one year.
  Consecutive sample (n=11) of adult patients requiring EVD placement, performed with AR guidance; compared to a matched (for quantity, intervention, performing surgeons, and timeframe), non-concurrent freehand control group (n=11, retrospective outcome analysis without active enrollment to receive study treatment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AR-assisted EVD placement (Experimental): External ventricular drain (EVD) placement using a standalone augmented reality (AR) headset equipped with high-accuracy inside-out infrared tracking and software addressing EVD placement.
  Interventions: Device: AR-assisted EVD placement; Procedure: Freehand EVD placement

INTERVENTIONS:
Device: AR-assisted EVD placement — Cfr. arm description
Procedure: Freehand EVD placement — External ventricular drain (EVD) placement using the conventional freehand technique. This intervention covers the matched, non-concurrent control group, retrospectively obtained without active enrollment to receive study treatment.

SUMMARY:
The goal of this clinical trial is to learn if high-accuracy augmented reality (AR) guidance for external ventricular drain (EVD) placement using a standalone head-worn navigation system can improve current shortcomings of freehand and image-guidance techniques. It will assess safety, feasibility and clinical performance. The main questions it aims to answer are:

* Is the implementation of a standalone head-worn AR navigation system for EVD placement in critical care settings feasible and safe?
* How does it compare to the conventional freehand technique in terms of EVD placement quality, complication rate and revision rate?

Researchers will assess placement quality using the modified Kakarla scale, grading placement quality based on the position of the EVD tip on postoperative CT imaging. The amount of attempts, complications and revisions will be documented. The results of the AR-guided placements will be compared to a matched, non-concurrent freehand control group.

Participants will undergo AR-guided EVD placement in a critical care setting (i.e. the emergency room or intensive care unit).

DETAILED DESCRIPTION:
External ventricular drain (EVD) placement is often performed using the freehand technique. In comparison to image-guided methods, this technique was identified as the primary risk factor of improper outcome, yielding optimal placement in only 70%. While conventional image guidance technologies introduce a distinct improvement in accuracy, these systems tend to be prohibitively large and lack mobility, restricting their use to the operating room. As such, their practical implementation in critical care settings is not always feasible due to time, availability, and cost constraints.

This study aims to address shortcomings in both conventional EVD placement and current image guidance technologies. To achieve this, first an AR headset-based navigation system was developed, providing high-accuracy inside-out infrared tracking and software features specifically focusing on EVD placement. Phantom studies were conducted, which proved successful, with a positive outcome of AR-guided EVD placement on phantom heads over the freehand technique. Given these results, the researchers aim to test the system in a clinical trial setting.

Given the additional layer of information on top of knowledge and experience regarding the freehand technique, it is hypothesized that AR guidance will result in an improved outcome, as was the case for conventional neuronavigation.

This study is a prospective clinical pilot study, with the goal to assess feasibility, safety and clinical performance of high-accuracy AR-guided EVD placement using a standalone head-worn navigation system in critical care settings at the Universitair Ziekenhuis Brussel over the course of one year. The outcome will be quantified using the modified Kakarla scale to assess EVD placement quality on postoperative CT imaging, as well as the amount of attempts, complications and revisions. The results of the AR-guided placements will be compared to a non-concurrent control group of matched (for quantity, intervention, performing surgeons and timeframe) freehand EVD placement cases that will be collected retrospectively.

The study protocol was approved by the Ethics Committee of the Universitair Ziekenhuis Brussel (ref. 2018/447) and validated by the Belgian Federal Agency of Medicines and Health Products (FAGG/AFMPS ref. 80M0764).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Indication for bedside EVD placement in a critical care setting (emergency room or intensive care unit) using a twistdrill
* EVD placement as sole cranial intervention

Exclusion Criteria:

* Other cranial intervention(s) expected within the first 24h after EVD placement
* EVD placement in the OR using a craniotome and/or conventional neuronavigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-29 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Clinical EVD placement quality | Within 24 hours after surgery
  External ventricular drain (EVD) placement quality assessment using the modified Kakarla scale (mKS; with grades I (a and b), II and III), grading placement quality based on the EVD tip position (identified on the postoperative CT imaging) from optimal placement (mKS grade Ia) to poor or failed placement (mKS grade III).

SECONDARY OUTCOMES:
Required attempts | During surgery
  The number of attempts required for successful ventricular puncture
Procedure-related complications | Within 7 days after surgery
  The amount and type of complications related to the EVD placement procedure (e.g. hemorrhage, infection)
Revision rate | Within 24 hours after surgery
  The amount of revisions required in case of non-functional EVD placement

OTHER OUTCOMES:
Subjective technology experience | Within 7 days after inclusion of the last patient
  All participating surgeons will be asked to complete a questionnaire gauging their subjective experience regarding the use of the system (likelihood of technology-acceptance cfr. UTAUT model, subjective ease-of-use, any discomforts)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data obtained through this study may be provided upon request to qualified researchers with academic interest in AR guidance for EVD placement. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party. For request approval and following investigator support, contact Dr. Frederick Van Gestel (frederick.vangestel@uzbrussel.be).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted after publication of a resulting manuscript. If approved, data will be made accessible for up to 12 months, with the possibility of extension considered on a case-by-case basis.
Access Criteria: Requests for IPD access can be submitted by qualified researchers pursuing academic or independent scientific research on AR guidance for EVD placement. Following review of the proposed data use (through a research proposal and SAP), approval may be granted after which a data sharing agreement will be set up. For more information or to submit a request, please contact Dr. Frederick Van Gestel (frederick.vangestel@uzbrussel.be).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT06571539/Prot_SAP_000.pdf